CLINICAL TRIAL: NCT04932616
Title: Use of the Functional Gait Assessment in Patients With Multiple Sclerosis: Examining Reliability Between Face-to-Face and Online Applications
Brief Title: Tele-Assessment and Face-to-Face Evaluation of Functional Gait Assessment in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Perim Zengin, Physiotherapist, Istanbul University - Cerrahpasa
Other Study IDs: 12015
Record Dates: First submitted 2021-06-06; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
Keywords: teleassessment; functional gait assessment; balance; walk
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Face To Face (Clinic) Group Functional Gait Assessment: Evaluations to be applied for the cultural adaptation and reliability study of the scale:
  Functional Gait Assessment, Timed Up and Go Test, Four-Step Square Test, Timed 25-Foot Walk Test, 12-Item Multiple Sclerosis Walking Scale Berg Balance Scale
- Tele- Assessment Group Functional Gait Assessment: The evaluation to be applied for the tele-evaluation reliability study of the scale:
  Functional Gait Assessment

SUMMARY:
The aim of the study is to examine the reliability of the method by applying the Functional Gait Assessment in patients with Multiple Sclerosis via online video conferencing. For this purpose, walking of each patient to be included in the study; The evaluation results will be compared and the intra-rater reliability will be investigated by evaluating both face-to-face and online video conferencing methods. Since the Functional Gait Assessment is not available in Turkish, the scale will also be validated by adapting it to Turkish within the scope of the study.

DETAILED DESCRIPTION:
As with all neurological diseases, it is important to use appropriate outcome measurements in the assessment of balance and gait disorders in patients with Multiple Sclerosis (MS), in order to determine the appropriate program for the patient in physiotherapy and rehabilitation applications, both face-to-face and through telerehabilitation. The scale recommended by a clinical practice guide developed with the support of the American Physiotherapy Association (APTA) and the Academy of Neurological Physiotherapy (ANPT) is the Functional Gait Assessment (FGA). According to this proposal, a Turkish version will be made within the scope of the study so that functional walking evaluation can be used in our country. A 2017 study on functional gait assessment and Multiple Sclerosis investigated the validity and sensitivity to changes in the original English version of the test in multiple sclerosis, and as a result, its validity was found for MS. Functional gait assessment does not have a reliability study for Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Having a definite diagnosis of MS of any clinical type according to the 2017 Mc Donalds criteria by a neurologist,
* 18 years and over
* Expanded Disability Status Scale (EDSS) score of 2,5-6
* Not having an attack within the last 30 days
* Voluntarily giving consent to participate in the study
* Absence of visual and auditory impairment for completion of assessments

For Tele-assessment:

* Having a walking area of at least 3 meters at home to evaluate walking
* Providing a care provider's supervision to ensure walking safety
* The patient or the caregiver can use the video conferencing software application from the phone or computer

Exclusion Criteria:

* Diagnosis of another neurological disease that affects the level of ambulation other than MS
* Receiving corticosteroid therapy within the last 1 month
* Limitation in range of motion of the lower extremities, which may affect standing and walking
* Pain that negatively affects walking in the lower extremity and lumbar area (etc., coxarthrosis, gonarthrosis, sciatica)
* Inability to stand up from a sitting position (Timed Up & Go Test requirement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis patients over the age of 18 who applied to the Memorial Sisli Hospital Neurology Outpatient Clinic and volunteered to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Functional Gait Assessment | change from baseline at 15 day
  The Functional Gait Assessment is a test designed to assess balance during various walking tasks. This test is a modification of the Dynamic Gait Index to increase reliability and reduce the ceiling effect. This test, which consists of 10 items, evaluates dynamic balance skills such as walking at normal and different speeds, walking with horizontal and vertical head movements, turning quickly, walking over objects, toe-heel walking, walking backwards, walking with eyes closed, and climbing stairs. Each item is scored between 0-3 points; 0 indicates that he is unable to perform that skill or severe gait or balance disorder is observed while performing that skill, and 3 indicates that he has achieved that skill normally. Points 1 and 2 are scored for each task separately for specific situations. Items are added to score the FGA and the maximum total score is set as 30.

SECONDARY OUTCOMES:
Timed 25-Foot Walk Test | Baseline
  It is a performance test that provides information about the participant's mobility and leg function. The standardized protocol is very simple. The participant will be requested to walk as quickly and safely as possible (ie maximum walking speed) along a clearly marked, linear 25 feet or 7.62 m track. The participant can use an assistive device while walking. The person will walk two different times on the marked track and the average of two consecutive attempts in seconds will be recorded as a result of the test.
Timed Up and Go Test | Baseline
  It is a test used to evaluate dynamic balance. The test measures the time it takes a participant to get up from the chair and walk 3 meters at a comfortable pace and return to the chair and sit down. The test begins when the participant gets up from the chair and ends when the participant sits down on the chair again. The time measured is recorded in seconds. A shorter period represents better mobility.
Berg Balance Test | Baseline
  It is a scale containing 14 instructions and a score of 0-4 is given by observing the patient's performance for each instruction. 0 points are given in cases where the patient cannot perform the activity at all, while 4 points are given when the patient completes the activity independently. The highest score is 56 and 0-20 points indicate balance disorder, 21-40 points indicate an acceptable balance, 41-56 points indicate the presence of a good balance. It takes between 10 and 20 minutes to complete the scale.
The Four Square Step Test | Baseline
  The Four Square Step Test (FSST) is used to assess dynamic stability and the ability of the subject to step over low objects forward, sideways, and backward.
12-item Multiple Sclerosis Walking Scale | Baseline
  The Multiple Sclerosis Walking Scale (MSWS-12) is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation. A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100. Walking improvement on the MSWS-12 is indicated by negative change scores.

CONTACTS AND LOCATIONS:
Overall Officials: Perim Zengin, M.Sc, Principal Investigator — Istanbul University-Cerrahpasa Institute of Postgraduate Education; Burcu Ersöz Hüseyinsinoğlu, Assoc. Prof., Study Chair — Istanbul University-Cerrahpasa Faculty of Health Science; Burcu Altunrende, Prof. Dr., Study Chair — Memorial Şişli Hospital, Neurology Clinic
Locations (1):
- Memorial Sisli Hospital, Neurology Clinic, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
A video recording of the Functional Gait Assessment conducted in the clinic for inter-rater reliability analysis will be shared.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Hatcher-Martin JM, Adams JL, Anderson ER, Bove R, Burrus TM, Chehrenama M, Dolan O'Brien M, Eliashiv DS, Erten-Lyons D, Giesser BS, Moo LR, Narayanaswami P, Rossi MA, Soni M, Tariq N, Tsao JW, Vargas BB, Vota SA, Wessels SR, Planalp H, Govindarajan R. Telemedicine in neurology: Telemedicine Work Group of the American Academy of Neurology update. Neurology. 2020 Jan 7;94(1):30-38. doi: 10.1212/WNL.0000000000008708. Epub 2019 Dec 4. PMID 31801829
- [Background] Forsberg A, Andreasson M, Nilsagard Y. The Functional Gait Assessment in People with Multiple Sclerosis: Validity and Sensitivity to Change. Int J MS Care. 2017 Mar-Apr;19(2):66-72. doi: 10.7224/1537-2073.2015-061. PMID 32607064
- [Background] Yeroushalmi S, Maloni H, Costello K, Wallin MT. Telemedicine and multiple sclerosis: A comprehensive literature review. J Telemed Telecare. 2020 Aug-Sep;26(7-8):400-413. doi: 10.1177/1357633X19840097. Epub 2019 May 1. PMID 31042118
- [Background] Khan F, Amatya B, Kesselring J, Galea M. Telerehabilitation for persons with multiple sclerosis. Cochrane Database Syst Rev. 2015 Apr 9;2015(4):CD010508. doi: 10.1002/14651858.CD010508.pub2. PMID 25854331
- [Background] Moore JL, Potter K, Blankshain K, Kaplan SL, O'Dwyer LC, Sullivan JE. A Core Set of Outcome Measures for Adults With Neurologic Conditions Undergoing Rehabilitation: A CLINICAL PRACTICE GUIDELINE. J Neurol Phys Ther. 2018 Jul;42(3):174-220. doi: 10.1097/NPT.0000000000000229. PMID 29901487
- [Background] Wrisley DM, Marchetti GF, Kuharsky DK, Whitney SL. Reliability, internal consistency, and validity of data obtained with the functional gait assessment. Phys Ther. 2004 Oct;84(10):906-18. PMID 15449976
- [Background] Kieseier BC, Pozzilli C. Assessing walking disability in multiple sclerosis. Mult Scler. 2012 Jul;18(7):914-24. doi: 10.1177/1352458512444498. Epub 2012 Apr 24. PMID 22740603
- [Background] Hobart JC, Riazi A, Lamping DL, Fitzpatrick R, Thompson AJ. Measuring the impact of MS on walking ability: the 12-Item MS Walking Scale (MSWS-12). Neurology. 2003 Jan 14;60(1):31-6. doi: 10.1212/wnl.60.1.31. PMID 12525714
- [Background] Motl RW, Snook EM. Confirmation and extension of the validity of the Multiple Sclerosis Walking Scale-12 (MSWS-12). J Neurol Sci. 2008 May 15;268(1-2):69-73. doi: 10.1016/j.jns.2007.11.003. Epub 2007 Dec 3. PMID 18061618
- [Background] Cattaneo D, Regola A, Meotti M. Validity of six balance disorders scales in persons with multiple sclerosis. Disabil Rehabil. 2006 Jun 30;28(12):789-95. doi: 10.1080/09638280500404289. PMID 16754576
- [Background] Kirkwood RN, Batista NCL, Marques LBF, de Melo Ocarino J, Neves LLA, de Souza Moreira B. Cross-cultural adaptation and reliability of the Functional Gait Assessment in older Brazilian adults. Braz J Phys Ther. 2021 Jan-Feb;25(1):78-85. doi: 10.1016/j.bjpt.2020.02.004. Epub 2020 Feb 28. PMID 32143957
- [Background] Weber, C., Schwieterman, M., Fier, K., Berni, J., Swartz, N., Phillips, R. S., & Reneker, J. C. (2016). Reliability and Validity of the Functional Gait Assessment: A Systematic Review. Physical & Occupational Therapy In Geriatrics, 34(1), 88-103.
- [Background] Forsberg A, Andreasson M, Nilsagard YE. Validity of the dynamic gait index in people with multiple sclerosis. Phys Ther. 2013 Oct;93(10):1369-76. doi: 10.2522/ptj.20120284. Epub 2013 May 2. PMID 23641026